CLINICAL TRIAL: NCT00092677
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Effects of Ezetimibe + Simvastatin on Clinical Outcomes in Patients With Aortic Stenosis
Brief Title: An Investigational Drug on Clinical Outcomes in Patients With Aortic Stenosis (Narrowing of the Major Blood Vessel of the Heart)(MK-0653A-043 AM4)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-043; 2004_050 (Other: Merck Study Number)
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Results first posted 2009-05-27 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- EZ/Simva 10/40 mg (Experimental): Ezetimibe 10 mg + Simvastatin 40 mg
  Interventions: Drug: ezetimibe (+) simvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: ezetimibe (+) simvastatin — Duration of Treatment: 4 years
  Other Names: MK0653A
  Arms: EZ/Simva 10/40 mg
Drug: Comparator: Placebo — matching Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether treatment with an investigational drug as compared to placebo will reduce the risk of major cardiovascular events in patients with aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45 to 85 with mild abnormalities of the aortic valve as confirmed by an echocardiogram.

Exclusion Criteria:

* Patients previously in a trial using the study drug, or currently taking any medications that are not allowed in this study.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1873 (Actual)
Dates: Start 2001-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossebo AB, Pedersen TR, Boman K, Brudi P, Chambers JB, Egstrup K, Gerdts E, Gohlke-Barwolf C, Holme I, Kesaniemi YA, Malbecq W, Nienaber CA, Ray S, Skjaerpe T, Wachtell K, Willenheimer R; SEAS Investigators. Intensive lipid lowering with simvastatin and ezetimibe in aortic stenosis. N Engl J Med. 2008 Sep 25;359(13):1343-56. doi: 10.1056/NEJMoa0804602. Epub 2008 Sep 2. PMID 18765433
- [Background] Steine K, Rossebo AB, Stugaard M, Pedersen TR. Left ventricular systolic and diastolic function in asymptomatic patients with moderate aortic stenosis. Am J Cardiol. 2008 Oct 1;102(7):897-901. doi: 10.1016/j.amjcard.2008.07.001. Epub 2008 Aug 26. PMID 18805118
- [Derived] Bahlmann E, Gerdts E, Einarsen E, Midtbo H, Pedersen ER, Rossebo A, Willems S, Cramariuc D. Impact of sex-specific thresholds for low flow in assessment of prognosis in concordantly and discordantly graded aortic valve stenosis. Eur Heart J Cardiovasc Imaging. 2025 Jan 31;26(2):280-286. doi: 10.1093/ehjci/jeae272. PMID 39467305
- [Derived] Hadziselimovic E, Greve AM, Sajadieh A, Olsen MH, Kesaniemi YA, Nienaber CA, Ray SG, Rossebo AB, Wachtell K, Nielsen OW. Association of high-sensitivity troponin T with outcomes in asymptomatic non-severe aortic stenosis: a post-hoc substudy of the SEAS trial. EClinicalMedicine. 2023 Feb 28;58:101875. doi: 10.1016/j.eclinm.2023.101875. eCollection 2023 Apr. PMID 36915288
- [Derived] Bahlmann E, Einarsen E, Cramariuc D, Pedersen ER, Rossebo AB, Midtbo H, Willems S, Gerdts E. Prognosis in asymptomatic patients with discordantly graded aortic valve stenosis based on pressure recovery adjusted valve area. Open Heart. 2022 Nov;9(2):e002159. doi: 10.1136/openhrt-2022-002159. PMID 36428084
- [Derived] Hadziselimovic E, Greve AM, Sajadieh A, Olsen MH, Kesaniemi YA, Nienaber CA, Ray SG, Rossebo AB, Willenheimer R, Wachtell K, Nielsen OW. Association of Annual N-Terminal Pro-Brain Natriuretic Peptide Measurements With Clinical Events in Patients With Asymptomatic Nonsevere Aortic Stenosis: A Post Hoc Substudy of the SEAS Trial. JAMA Cardiol. 2022 Apr 1;7(4):435-444. doi: 10.1001/jamacardio.2021.5916. PMID 35171199
- [Derived] Bahlmann E, Einarsen E, Cramariuc D, Midtbo H, Mancusi C, Rossebo A, Willems S, Gerdts E. Low myocardial energetic efficiency is associated with increased mortality in aortic stenosis. Open Heart. 2021 Aug;8(2):e001720. doi: 10.1136/openhrt-2021-001720. PMID 34426527
- [Derived] Einarsen E, Cramariuc D, Bahlmann E, Midtbo H, Chambers JB, Gerdts E. Higher Acceleration/Ejection Time Ratio Predicts Impaired Outcome in Aortic Valve Stenosis. Circ Cardiovasc Imaging. 2021 Jan;14(1):e011467. doi: 10.1161/CIRCIMAGING.120.011467. Epub 2021 Jan 19. PMID 33461302
- [Derived] Greve AM, Bang CN, Boman K, Egstrup K, Kesaniemi YA, Ray S, Pedersen TR, Wachtell K. Relation of Lipid-Lowering Therapy to Need for Aortic Valve Replacement in Patients With Asymptomatic Mild to Moderate Aortic Stenosis. Am J Cardiol. 2019 Dec 1;124(11):1736-1740. doi: 10.1016/j.amjcard.2019.08.037. Epub 2019 Sep 7. PMID 31586530
- [Derived] Gerdts E, Saeed S, Midtbo H, Rossebo A, Chambers JB, Einarsen E, Bahlmann E, Devereux R. Higher left ventricular mass-wall stress-heart rate product and outcome in aortic valve stenosis. Heart. 2019 Nov;105(21):1629-1633. doi: 10.1136/heartjnl-2018-314462. Epub 2019 Jun 1. PMID 31154431
- [Derived] Bahlmann E, Cramariuc D, Saeed S, Chambers JB, Nienaber CA, Kuck KH, Lonnebakken MT, Gerdts E. Low systemic arterial compliance is associated with increased cardiovascular morbidity and mortality in aortic valve stenosis. Heart. 2019 Oct;105(19):1507-1514. doi: 10.1136/heartjnl-2018-314386. Epub 2019 May 15. PMID 31092548
- [Derived] Hodges GW, Bang CN, Forman JL, Olsen MH, Boman K, Ray S, Kesaniemi YA, Eugen-Olsen J, Greve AM, Jeppesen JL, Wachtell K. Effect of simvastatin and ezetimibe on suPAR levels and outcomes. Atherosclerosis. 2018 May;272:129-136. doi: 10.1016/j.atherosclerosis.2018.03.030. Epub 2018 Mar 16. PMID 29602140
- [Derived] Hodges GW, Bang CN, Eugen-Olsen J, Olsen MH, Boman K, Ray S, Kesaniemi AY, Jeppesen JL, Wachtell K. SuPAR predicts postoperative complications and mortality in patients with asymptomatic aortic stenosis. Open Heart. 2018 Jan 13;5(1):e000743. doi: 10.1136/openhrt-2017-000743. eCollection 2018. PMID 29387432
- [Derived] Greve AM, Bang CN, Boman K, Egstrup K, Forman JL, Kesaniemi YA, Ray S, Pedersen TR, Best P, Rajamannan NM, Wachtell K. Effect Modifications of Lipid-Lowering Therapy on Progression of Aortic Stenosis (from the Simvastatin and Ezetimibe in Aortic Stenosis [SEAS] Study). Am J Cardiol. 2018 Mar 15;121(6):739-745. doi: 10.1016/j.amjcard.2017.12.011. Epub 2017 Dec 25. PMID 29361285
- [Derived] Bang CN, Greve AM, Rossebo AB, Ray S, Egstrup K, Boman K, Nienaber C, Okin PM, Devereux RB, Wachtell K. Antihypertensive Treatment With beta-Blockade in Patients With Asymptomatic Aortic Stenosis and Association With Cardiovascular Events. J Am Heart Assoc. 2017 Nov 27;6(12):e006709. doi: 10.1161/JAHA.117.006709. PMID 29180457
- [Derived] Saeed S, Senior R, Chahal NS, Lonnebakken MT, Chambers JB, Bahlmann E, Gerdts E. Lower Transaortic Flow Rate Is Associated With Increased Mortality in Aortic Valve Stenosis. JACC Cardiovasc Imaging. 2017 Aug;10(8):912-920. doi: 10.1016/j.jcmg.2017.05.008. PMID 28797414
- [Derived] Thomassen HK, Cioffi G, Gerdts E, Einarsen E, Midtbo HB, Mancusi C, Cramariuc D. Echocardiographic aortic valve calcification and outcomes in women and men with aortic stenosis. Heart. 2017 Oct;103(20):1619-1624. doi: 10.1136/heartjnl-2016-311040. Epub 2017 Jul 11. PMID 28698175
- [Derived] Lonnebakken MT, De Simone G, Saeed S, Boman K, Rossebo AB, Bahlmann E, Gohlke-Barwolf C, Gerdts E. Impact of stroke volume on cardiovascular risk during progression of aortic valve stenosis. Heart. 2017 Sep;103(18):1443-1448. doi: 10.1136/heartjnl-2016-310917. Epub 2017 Apr 28. PMID 28455295
- [Derived] Bahlmann E, Cramariuc D, Minners J, Lonnebakken MT, Ray S, Gohlke-Baerwolf C, Nienaber CA, Jander N, Seifert R, Chambers JB, Kuck KH, Gerdts E. Small aortic root in aortic valve stenosis: clinical characteristics and prognostic implications. Eur Heart J Cardiovasc Imaging. 2017 Apr 1;18(4):404-412. doi: 10.1093/ehjci/jew159. PMID 27491438
- [Derived] Nielsen OW, Sajadieh A, Sabbah M, Greve AM, Olsen MH, Boman K, Nienaber CA, Kesaniemi YA, Pedersen TR, Willenheimer R, Wachtell K. Assessing Optimal Blood Pressure in Patients With Asymptomatic Aortic Valve Stenosis: The Simvastatin Ezetimibe in Aortic Stenosis Study (SEAS). Circulation. 2016 Aug 9;134(6):455-68. doi: 10.1161/CIRCULATIONAHA.115.021213. Epub 2016 Aug 2. PMID 27486164
- [Derived] Bang CN, Greve AM, La Cour M, Boman K, Gohlke-Barwolf C, Ray S, Pedersen T, Rossebo A, Okin PM, Devereux RB, Wachtell K. Effect of Randomized Lipid Lowering With Simvastatin and Ezetimibe on Cataract Development (from the Simvastatin and Ezetimibe in Aortic Stenosis Study). Am J Cardiol. 2015 Dec 15;116(12):1840-4. doi: 10.1016/j.amjcard.2015.09.026. Epub 2015 Oct 3. PMID 26602073
- [Derived] Gerdts E, Rossebo AB, Pedersen TR, Cioffi G, Lonnebakken MT, Cramariuc D, Rogge BP, Devereux RB. Relation of Left Ventricular Mass to Prognosis in Initially Asymptomatic Mild to Moderate Aortic Valve Stenosis. Circ Cardiovasc Imaging. 2015 Nov;8(11):e003644; discussion e003644. doi: 10.1161/CIRCIMAGING.115.003644. PMID 26489804
- [Derived] Blyme A, Asferg C, Nielsen OW, Sehestedt T, Kesaniemi YA, Gohlke-Barwolf C, Boman K, Willenheimer R, Ray S, Nienaber CA, Rossebo A, Wachtell K, Olsen MH. High sensitivity C reactive protein as a prognostic marker in patients with mild to moderate aortic valve stenosis during lipid-lowering treatment: an SEAS substudy. Open Heart. 2015 Feb 4;2(1):e000152. doi: 10.1136/openhrt-2014-000152. eCollection 2015. PMID 25685360
- [Derived] Greve AM, Bang CN, Berg RM, Egstrup K, Rossebo AB, Boman K, Nienaber CA, Ray S, Gohlke-Baerwolf C, Nielsen OW, Okin PM, Devereux RB, Kober L, Wachtell K. Resting heart rate and risk of adverse cardiovascular outcomes in asymptomatic aortic stenosis: the SEAS study. Int J Cardiol. 2015 Feb 1;180:122-8. doi: 10.1016/j.ijcard.2014.11.181. Epub 2014 Nov 26. PMID 25438232
- [Derived] Cramariuc D, Rogge BP, Lonnebakken MT, Boman K, Bahlmann E, Gohlke-Barwolf C, Chambers JB, Pedersen TR, Gerdts E. Sex differences in cardiovascular outcome during progression of aortic valve stenosis. Heart. 2015 Feb;101(3):209-14. doi: 10.1136/heartjnl-2014-306078. Epub 2014 Oct 9. PMID 25301859
- [Derived] Jander N, Hochholzer W, Kaufmann BA, Bahlmann E, Gerdts E, Boman K, Chambers JB, Nienaber CA, Ray S, Rossebo A, Pedersen TR, Wachtell K, Gohlke-Barwolf C, Neumann FJ, Minners J. Velocity ratio predicts outcomes in patients with low gradient severe aortic stenosis and preserved EF. Heart. 2014 Dec;100(24):1946-53. doi: 10.1136/heartjnl-2014-305763. Epub 2014 Sep 12. PMID 25217488
- [Derived] Greve AM, Dalsgaard M, Bang CN, Egstrup K, Rossebo AB, Boman K, Cramariuc D, Nienaber CA, Ray S, Gohlke-Baerwolf C, Okin PM, Devereux RB, Kober L, Wachtell K. Usefulness of the electrocardiogram in predicting cardiovascular mortality in asymptomatic adults with aortic stenosis (from the Simvastatin and Ezetimibe in Aortic Stenosis Study). Am J Cardiol. 2014 Sep 1;114(5):751-6. doi: 10.1016/j.amjcard.2014.06.006. Epub 2014 Jun 21. PMID 25048345
- [Derived] Greve AM, Dalsgaard M, Bang CN, Egstrup K, Ray S, Boman K, Rossebo AB, Gohlke-Baerwolf C, Devereux RB, Kober L, Wachtell K. Stroke in patients with aortic stenosis: the Simvastatin and Ezetimibe in Aortic Stenosis study. Stroke. 2014 Jul;45(7):1939-46. doi: 10.1161/STROKEAHA.114.005296. Epub 2014 Jun 5. PMID 24903982
- [Derived] Minners J, Gohlke-Baerwolf C, Kaufmann BA, Bahlmann E, Gerdts E, Boman K, Chambers JB, Nienaber CA, Willenheimer R, Wachtell K, Holme I, Pedersen TR, Neumann FJ, Jander N. Adjusting parameters of aortic valve stenosis severity by body size. Heart. 2014 Jul;100(13):1024-30. doi: 10.1136/heartjnl-2013-305225. Epub 2014 Apr 29. PMID 24780909
- [Derived] Bahlmann E, Gerdts E, Cramariuc D, Gohlke-Baerwolf C, Nienaber CA, Wachtell K, Seifert R, Chambers JB, Kuck KH, Ray S. Prognostic value of energy loss index in asymptomatic aortic stenosis. Circulation. 2013 Mar 12;127(10):1149-56. doi: 10.1161/CIRCULATIONAHA.112.078857. Epub 2013 Jan 28. PMID 23357717
- [Derived] Greve AM, Gerdts E, Boman K, Gohlke-Baerwolf C, Rossebo AB, Devereux RB, Kober L, Ray S, Willenheimer R, Wachtell K. Impact of QRS duration and morphology on the risk of sudden cardiac death in asymptomatic patients with aortic stenosis: the SEAS (Simvastatin and Ezetimibe in Aortic Stenosis) Study. J Am Coll Cardiol. 2012 Mar 27;59(13):1142-9. doi: 10.1016/j.jacc.2011.12.020. PMID 22440214
- [Derived] Holme I, Pedersen TR, Boman K, Egstrup K, Gerdts E, Kesaniemi YA, Malbecq W, Ray S, Rossebo AB, Wachtell K, Willenheimer R, Gohlke-Barwolf C. A risk score for predicting mortality in patients with asymptomatic mild to moderate aortic stenosis. Heart. 2012 Mar;98(5):377-83. doi: 10.1136/heartjnl-2011-300475. Epub 2011 Dec 8. PMID 22155702
- [Derived] Greve AM, Boman K, Gohlke-Baerwolf C, Kesaniemi YA, Nienaber C, Ray S, Egstrup K, Rossebo AB, Devereux RB, Kober L, Willenheimer R, Wachtell K. Clinical implications of electrocardiographic left ventricular strain and hypertrophy in asymptomatic patients with aortic stenosis: the Simvastatin and Ezetimibe in Aortic Stenosis study. Circulation. 2012 Jan 17;125(2):346-53. doi: 10.1161/CIRCULATIONAHA.111.049759. Epub 2011 Dec 6. PMID 22147903
- [Derived] Cramariuc D, Cioffi G, Rieck AE, Devereux RB, Staal EM, Ray S, Wachtell K, Gerdts E. Low-flow aortic stenosis in asymptomatic patients: valvular-arterial impedance and systolic function from the SEAS Substudy. JACC Cardiovasc Imaging. 2009 Apr;2(4):390-9. doi: 10.1016/j.jcmg.2008.12.021. PMID 19580719
- [Derived] Peto R, Emberson J, Landray M, Baigent C, Collins R, Clare R, Califf R. Analyses of cancer data from three ezetimibe trials. N Engl J Med. 2008 Sep 25;359(13):1357-66. doi: 10.1056/NEJMsa0806603. Epub 2008 Sep 2. PMID 18765432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III. Study Initiation Date (FPI) was 06-Jan-2003 and Study Completion Date (LPO) was 17-Apr-2008. Primary therapy period 02-Mar-2001 to 31-Mar-2008 includes start date of therapy from the Simvastatin in Aortic Stenosis (SAS) study. 173 study centers worldwide (Denmark, Finland, Germany, Great Britain, Ireland, Norway, and Sweden)
Pre-assignment Details: Included patients with asymptomatic aortic stenosis as assessed on echocardiography, not requiring lipid-lowering therapy, and without known coronary heart disease or diabetes mellitus. 4 week placebo/diet run-in period was followed by treatment period lasting until 4 years after the last patient was randomized.
Period: Overall Study
Arm/Group | EZ/Simva 10/40 mg | Placebo
Started | 944 | 929
Completed | 939 (EZ/Simva: 694 (on drug), 140 (after drug discon), 105 (at death)) | 918 (Placebo: 698 (on drug), 120 (after drug discon), 100 (at death))
Not Completed | 5 | 11
Not completed — Lost to Follow-up | 0 | 2
Not completed — Adminstrative | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EZ/Simva 10/40 mg | Placebo | Total
Number analyzed (Participants) | 944 | 929 | 1873
Age, Continuous [Mean (Full Range); unit: years] | 67.7 [41 to 86] | 67.4 [28 to 85] | 67.5 [28 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 363 | 360 | 723
  Male | 581 | 569 | 1150
Race/Ethnicity, Customized [Number; unit: participants]
  White | 940 | 928 | 1868
  Asian | 3 | 1 | 4
  Other | 1 | 0 | 1
High-density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mmol/L] | 1.49 (0.43) | 1.49 (0.43) | 1.49 (0.43)
Low-density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mmol/L] | 3.62 (0.93) | 3.59 (0.91) | 3.60 (0.92)
Peak Transaortic Jet Velocity [Mean (Standard Deviation); unit: m/sec] | 3.09 (0.55) | 3.10 (0.54) | 3.09 (0.54)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.76 (1.04) | 5.73 (0.99) | 5.74 (1.02)
Triglycerides (TG) [Mean (Standard Deviation); unit: mmol/L] | 1.42 (0.71) | 1.42 (0.68) | 1.42 (0.69)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced One or More Components of the Composite Clinical Endpoint of MCE (Major Cardiovascular Events)
Description: Composite endpoint of MCE consists of cardiovascular death, AVR (aortic valve replacement) surgery, CHF(congestive heart failure) as a result of progression of aortic stenosis, nonfatal MI (myocardial infarction), CABG (coronary artery bypass) surgery, PCI (percutaneous coronary intervention), hospitalized unstable angina, and nonhemorrhagic stroke
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 333 | 355
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.591, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 0.960, 95% CI [0.826 to 1.115] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

2. Secondary Outcome: Number of Participants That Experienced One or More Components of the Composite Clinical Endpoint of AVE (Aortic Valve Events)
Description: Composite endpoint of AVE (aortic valve events) consists of AVR surgery, CHF (as a result of progression of AS), or cardiovascular death
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 308 | 326
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.732, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 0.973, 95% CI [0.833 to 1.137] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

3. Secondary Outcome: Number of Participants That Experienced One or More Components of the Composite Clinical Endpoint of ICE (Ischemic Cardiovascular Events)
Description: Composite endpoint of ICE (ischemic cardiovascular events) consists of cardiovascular death, nonfatal MI, CABG, PCI, hospitalized unstable angina, and nonhemorrhagic stroke
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 148 | 187
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.024, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 0.780, 95% CI [0.628 to 0.967] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

4. Other Pre Specified Outcome: Cardiovascular Death
Description: Number of participants that experienced cardiovascular death
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 47 | 56
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.344, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 0.829, 95% CI [0.563 to 1.222] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

5. Other Pre Specified Outcome: Aortic Valve Replacement (AVR)
Description: Number of participants that experienced aortic valve replacement (AVR)
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 267 | 278
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.968, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 0.997, 95% CI [0.842 to 1.179] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

6. Other Pre Specified Outcome: Congestive Heart Failure (CHF) Due to Progression of Aortic Stenosis (AS)
Description: Number of participants that experienced Congestive Heart Failure (CHF) due to progression of aortic stenosis (AS)
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 25 | 23
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.771, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 1.088, 95% CI [0.617 to 1.917] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

7. Other Pre Specified Outcome: Nonfatal Myocardial Infarction (MI)
Description: Number of participants that experienced nonfatal myocardial infarction (MI)
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 17 | 26
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.147, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 0.636, 95% CI [0.345 to 1.173] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

8. Other Pre Specified Outcome: Coronary Artery Bypass Grafting (CABG)
Description: Number of participants that experienced coronary artery bypass grafting (CABG)
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 69 | 100
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.015, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 0.683, 95% CI [0.503 to 0.929] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

9. Other Pre Specified Outcome: Percutaneous Coronary Intervention (PCI)
Description: Number of participants that experienced percutaneous coronary intervention (PCI)
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 8 | 17
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; Regression, Cox — The p-value was not provided as there were less than 40 patients who reported the specific endpoint; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 0.456, 95% CI [0.197 to 1.057] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

10. Other Pre Specified Outcome: Hospitalization for Unstable Angina
Description: Number of participants that experienced hospitalization for unstable angina
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 5 | 8
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; Regression, Cox — The p-value was not provided as there were less than 40 patients who reported the specific endpoint; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 0.608, 95% CI [0.199 to 1.860] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

11. Other Pre Specified Outcome: Nonhemorrhagic Stroke
Description: Number of participants that experienced nonhemorrhagic stroke
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 33 | 29
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.647, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 1.124, 95% CI [0.682 to 1.850] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

12. Other Pre Specified Outcome: Death (Any Cause)
Description: Number of participants that died (any cause)
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 105 | 100
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.799, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 1.036, 95% CI [0.788 to 1.363] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

13. Post Hoc Outcome: Death Due to Cancer
Description: Number of participants that died due to cancer
Time Frame: Entire follow-up (median = 4.35 years)
Population: Intention-to-Treat
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 944 | 929
Participants | 39 | 23
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.052, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 1.667, 95% CI [0.996 to 2.791] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

14. Post Hoc Outcome: Incident Cancer
Description: Number of participants with incident cancer
Time Frame: Entire follow-up (median = 4.35 years)
Population: One patient from the 944 patients randomized to ezetimibe/simvastatin 10/40 mg did not receive study medication and was not included.
Measure: Number; unit: Participants
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 943 | 929
Participants | 105 | 70
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.008, Regression, Cox; Model terms: treatment and baseline peak transaortic jet velocity (as continuous covariate); Hazard Ratio (HR) = 1.504, 95% CI [1.111 to 2.035] — Direction of the Comparison: Hazard Ratio of experiencing the endpoint on EZ/Simva 10/40 mg compared to Placebo

15. Secondary Outcome: Change From Baseline in Peak Transaortic Jet Velocity
Description: Mean change from baseline in peak transaortic jet velocity
Time Frame: Baseline to End of follow-up (median = 4.35 years) or pre-aortic valve replacement
Population: Full Analysis Set: All patients who were randomized, took at least one dose of blinded study therapy and had a baseline and at least one post-randomization assessment without regard to protocol violations or compliance with study medication. 180 patients were excluded from peak transaortic jet velocity due to missing measurements.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 859 | 834
m/sec | 0.613 (0.586) | 0.618 (0.612)
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p = 0.829, ANCOVA; Model terms: treatment and baseline peak transaortic jet velocity; Mean Difference (Final Values) = -0.006, 95% CI [-0.063 to 0.051], Standard Error of Mean 0.029 — Direction of the Comparison: EZ/Simva 10/40 mg minus Placebo

16. Other Pre Specified Outcome: Percent Change in Time Weighted Average Total Cholesterol From Baseline to End of Follow-up
Description: Mean percent change (time-weighted average over follow-up) from baseline: Time-weighted average calculated using values at week 8, week 24, year 1 and every 6 months with time interval (days) between 2 successive values used as the weighting factor. For the first follow-up value, the weight was the number of days from randomization.
Time Frame: Baseline to End of follow-up (median = 4.35 years)
Population: Full Analysis Set: All patients who were randomized, took at least one dose of blinded study therapy and had a baseline and at least one post-randomization assessment without regard to protocol violations or compliance with study medication.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 937 | 916
Percent Change | -34.8 (13.5) | -2.7 (11.8)
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p <= 0.001, ANOVA; Model terms: treatment; Mean Difference (Final Values) = -32.1, 95% CI [-33.3 to -31.0], Standard Error of Mean 0.6 — Direction of the Comparison: EZ/Simva 10/40 mg minus Placebo

17. Other Pre Specified Outcome: Percent Change in Time Weighted Average Low-density Lipoprotein Cholesterol (LDL-C) From Baseline to End of Follow-up
Description: as for outcome 16
Time Frame: Baseline to End of follow-up (median = 4.35 years)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 937 | 916
Percent Change | -53.8 (18.7) | -3.8 (20.6)
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p <= 0.001, ANOVA; Model terms: treatment; Mean Difference (Final Values) = -50.0, 95% CI [-51.8 to -48.2], Standard Error of Mean 0.9 — Direction of the Comparison: EZ/Simva 10/40 mg minus Placebo

18. Other Pre Specified Outcome: Percent Change in Time Weighted Average High-density Lipoprotein Cholesterol (HDL-C) From Baseline to End of Follow-up
Description: as for outcome 16
Time Frame: Baseline to End of follow-up (median = 4.35 years)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 937 | 916
Percent change | 6.5 (17.7) | 2.5 (16.1)
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p <= 0.001, ANOVA; Model terms: treatment; Mean Difference (Final Values) = 3.9, 95% CI [2.4 to 5.5], Standard Error of Mean 0.8 — Direction of the Comparison: EZ/Simva 10/40 mg minus Placebo

19. Other Pre Specified Outcome: Percent Change in Time Weighted Average Triglycerides From Baseline to End of Follow-up
Description: as for outcome 16
Time Frame: Baseline to End of follow-up (median = 4.35 years)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | EZ/Simva 10/40 mg | Placebo
Number analyzed (Participants) | 937 | 916
Percent Change | -14.9 (27.6) | 5.1 (30.4)
Statistical Analysis 1: Comparison: EZ/Simva 10/40 mg vs Placebo; Test type: Superiority or Other; p <= 0.001, ANOVA; Model terms: treatment; Mean Difference (Final Values) = -20.0, 95% CI [-22.6 to -17.3], Standard Error of Mean 1.3 — Direction of the Comparison: EZ/Simva 10/40 mg minus Placebo

ADVERSE EVENTS:
Arm/Group | EZ/Simva 10/40 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 471 | 465
Other Adverse Events (participants affected / at risk) | 703 | 706
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | EZ/Simva 10/40 mg | Placebo
Anaemia (Blood and lymphatic system disorders) | 12/943 | 8/929
Haemolytic anaemia (Blood and lymphatic system disorders) | 1/943 | 0/929
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1/943 | 2/929
Pernicious anaemia (Blood and lymphatic system disorders) | 0/943 | 1/929
AV dissociation (Cardiac disorders) | 0/943 | 1/929
Acute coronary syndrome (Cardiac disorders) | 0/943 | 2/929
Acute myocardial infarction (Cardiac disorders) | 2/943 | 0/929
Angina pectoris (Cardiac disorders) | 3/943 | 8/929
Aortic valve disease mixed (Cardiac disorders) | 0/943 | 1/929
Aortic valve incompetence (Cardiac disorders) | 1/943 | 1/929
Aortic valve stenosis (Cardiac disorders) | 69/943 | 60/929
Arrhythmia (Cardiac disorders) | 2/943 | 2/929
Arteriosclerosis coronary artery (Cardiac disorders) | 0/943 | 1/929
Atrial fibrillation (Cardiac disorders) | 45/943 | 27/929
Atrial flutter (Cardiac disorders) | 8/943 | 1/929
Atrial tachycardia (Cardiac disorders) | 1/943 | 0/929
Atrial thrombosis (Cardiac disorders) | 0/943 | 1/929
Atrioventricular block (Cardiac disorders) | 2/943 | 2/929
Atrioventricular block complete (Cardiac disorders) | 6/943 | 5/929
Atrioventricular block second degree (Cardiac disorders) | 1/943 | 3/929
Bradyarrhythmia (Cardiac disorders) | 2/943 | 0/929
Bradycardia (Cardiac disorders) | 0/943 | 1/929
Cardiac amyloidosis (Cardiac disorders) | 0/943 | 1/929
Cardiac arrest (Cardiac disorders) | 2/943 | 1/929
Cardiac disorder (Cardiac disorders) | 0/943 | 1/929
Cardiac failure (Cardiac disorders) | 5/943 | 6/929
Cardiac failure acute (Cardiac disorders) | 1/943 | 1/929
Cardiac failure congestive (Cardiac disorders) | 1/943 | 1/929
Cardiac tamponade (Cardiac disorders) | 1/943 | 0/929
Cardiovascular disorder (Cardiac disorders) | 1/943 | 0/929
Coronary artery disease (Cardiac disorders) | 2/943 | 5/929
Coronary artery stenosis (Cardiac disorders) | 2/943 | 0/929
Dressler's syndrome (Cardiac disorders) | 1/943 | 0/929
Extrasystoles (Cardiac disorders) | 1/943 | 0/929
Hypertrophic cardiomyopathy (Cardiac disorders) | 1/943 | 0/929
Myocardial infarction (Cardiac disorders) | 7/943 | 7/929
Myocardial ischaemia (Cardiac disorders) | 3/943 | 0/929
Myocarditis (Cardiac disorders) | 1/943 | 0/929
Nodal arrhythmia (Cardiac disorders) | 0/943 | 1/929
Palpitations (Cardiac disorders) | 2/943 | 3/929
Pericardial effusion (Cardiac disorders) | 5/943 | 7/929
Pericardial haemorrhage (Cardiac disorders) | 1/943 | 1/929
Sick sinus syndrome (Cardiac disorders) | 4/943 | 6/929
Silent myocardial infarction (Cardiac disorders) | 1/943 | 0/929
Sinoatrial block (Cardiac disorders) | 2/943 | 0/929
Supraventricular tachycardia (Cardiac disorders) | 2/943 | 1/929
Tachyarrhythmia (Cardiac disorders) | 1/943 | 0/929
Tachycardia (Cardiac disorders) | 1/943 | 0/929
Tachycardia paroxysmal (Cardiac disorders) | 1/943 | 0/929
Ventricular arrhythmia (Cardiac disorders) | 0/943 | 1/929
Ventricular extrasystoles (Cardiac disorders) | 1/943 | 0/929
Ventricular fibrillation (Cardiac disorders) | 3/943 | 1/929
Ventricular tachycardia (Cardiac disorders) | 1/943 | 1/929
Dermoid cyst (Congenital, familial and genetic disorders) | 1/943 | 0/929
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 1/943 | 1/929
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 1/943 | 1/929
Hydrocele (Congenital, familial and genetic disorders) | 1/943 | 0/929
Phimosis (Congenital, familial and genetic disorders) | 0/943 | 1/929
Deafness neurosensory (Ear and labyrinth disorders) | 0/943 | 1/929
Deafness unilateral (Ear and labyrinth disorders) | 1/943 | 0/929
Vertigo (Ear and labyrinth disorders) | 6/943 | 7/929
Goitre (Endocrine disorders) | 0/943 | 2/929
Hyperthyroidism (Endocrine disorders) | 2/943 | 0/929
Amaurosis fugax (Eye disorders) | 0/943 | 1/929
Cataract (Eye disorders) | 3/943 | 6/929
Dacryostenosis acquired (Eye disorders) | 0/943 | 1/929
Diplopia (Eye disorders) | 0/943 | 1/929
Eye haemorrhage (Eye disorders) | 0/943 | 1/929
Glaucoma (Eye disorders) | 1/943 | 3/929
Retinal artery occlusion (Eye disorders) | 3/943 | 1/929
Retinal detachment (Eye disorders) | 2/943 | 2/929
Vitreous haemorrhage (Eye disorders) | 0/943 | 1/929
Abdominal discomfort (Gastrointestinal disorders) | 1/943 | 0/929
Abdominal hernia (Gastrointestinal disorders) | 0/943 | 2/929
Abdominal pain (Gastrointestinal disorders) | 9/943 | 5/929
Abdominal pain upper (Gastrointestinal disorders) | 0/943 | 3/929
Anal polyp (Gastrointestinal disorders) | 1/943 | 0/929
Anal stenosis (Gastrointestinal disorders) | 0/943 | 1/929
Appendicitis perforated (Gastrointestinal disorders) | 1/943 | 1/929
Colitis ischaemic (Gastrointestinal disorders) | 0/943 | 1/929
Colonic obstruction (Gastrointestinal disorders) | 1/943 | 0/929
Constipation (Gastrointestinal disorders) | 3/943 | 2/929
Crohn's disease (Gastrointestinal disorders) | 1/943 | 1/929
Diarrhoea (Gastrointestinal disorders) | 0/943 | 2/929
Diverticulum (Gastrointestinal disorders) | 1/943 | 0/929
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1/943 | 0/929
Duodenal ulcer (Gastrointestinal disorders) | 3/943 | 3/929
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1/943 | 0/929
Dyspepsia (Gastrointestinal disorders) | 1/943 | 2/929
Dysphagia (Gastrointestinal disorders) | 1/943 | 0/929
Faecal incontinence (Gastrointestinal disorders) | 0/943 | 1/929
Gastric haemorrhage (Gastrointestinal disorders) | 0/943 | 1/929
Gastric ulcer (Gastrointestinal disorders) | 7/943 | 2/929
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1/943 | 0/929
Gastritis (Gastrointestinal disorders) | 1/943 | 1/929
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/943 | 3/929
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2/943 | 0/929
Haematemesis (Gastrointestinal disorders) | 1/943 | 0/929
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1/943 | 2/929
Haemorrhoids (Gastrointestinal disorders) | 0/943 | 2/929
Heyde's syndrome (Gastrointestinal disorders) | 1/943 | 0/929
Hiatus hernia (Gastrointestinal disorders) | 1/943 | 1/929
Ileus (Gastrointestinal disorders) | 2/943 | 0/929
Ileus paralytic (Gastrointestinal disorders) | 1/943 | 1/929
Inguinal hernia (Gastrointestinal disorders) | 15/943 | 15/929
Intestinal ulcer (Gastrointestinal disorders) | 0/943 | 1/929
Large intestinal ulcer (Gastrointestinal disorders) | 1/943 | 0/929
Mechanical ileus (Gastrointestinal disorders) | 2/943 | 0/929
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1/943 | 0/929
Mouth haemorrhage (Gastrointestinal disorders) | 0/943 | 1/929
Nausea (Gastrointestinal disorders) | 2/943 | 5/929
Necrotising oesophagitis (Gastrointestinal disorders) | 0/943 | 1/929
Oesophagitis (Gastrointestinal disorders) | 0/943 | 2/929
Pancreatitis (Gastrointestinal disorders) | 2/943 | 1/929
Pancreatitis acute (Gastrointestinal disorders) | 0/943 | 1/929
Peptic ulcer (Gastrointestinal disorders) | 1/943 | 0/929
Peritonitis (Gastrointestinal disorders) | 2/943 | 0/929
Rectal haemorrhage (Gastrointestinal disorders) | 4/943 | 1/929
Reflux oesophagitis (Gastrointestinal disorders) | 0/943 | 1/929
Retroperitoneal haematoma (Gastrointestinal disorders) | 0/943 | 1/929
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1/943 | 0/929
Umbilical hernia (Gastrointestinal disorders) | 1/943 | 2/929
Vomiting (Gastrointestinal disorders) | 2/943 | 0/929
Alanine aminotransferase increased (General disorders) | 2/943 | 0/929
Aspartate aminotransferase increased (General disorders) | 3/943 | 0/929
Blood creatine phosphokinase increased (General disorders) | 1/943 | 0/929
Blood creatinine increased (General disorders) | 1/943 | 0/929
Blood potassium increased (General disorders) | 1/943 | 0/929
Blood sodium decreased (General disorders) | 1/943 | 0/929
Blood urine present (General disorders) | 0/943 | 1/929
C-reactive protein increased (General disorders) | 0/943 | 1/929
Cardiac output decreased (General disorders) | 0/943 | 1/929
Ejection fraction decreased (General disorders) | 1/943 | 1/929
Electrocardiogram abnormal (General disorders) | 2/943 | 0/929
Haemoglobin decreased (General disorders) | 0/943 | 1/929
International normalised ratio (General disorders) | 1/943 | 0/929
International normalised ratio decreased (General disorders) | 1/943 | 0/929
International normalised ratio increased (General disorders) | 3/943 | 4/929
Occult blood positive (General disorders) | 0/943 | 1/929
Platelet count decreased (General disorders) | 1/943 | 1/929
Prostatic specific antigen increased (General disorders) | 1/943 | 0/929
Pulmonary function test decreased (General disorders) | 0/943 | 1/929
Total lung capacity decreased (General disorders) | 0/943 | 1/929
Weight decreased (General disorders) | 1/943 | 1/929
Adverse drug reaction (General disorders) | 1/943 | 0/929
Asthenia (General disorders) | 1/943 | 0/929
Atrophy (General disorders) | 0/943 | 1/929
Catheter related complication (General disorders) | 1/943 | 1/929
Catheter site haemorrhage (General disorders) | 1/943 | 0/929
Chest discomfort (General disorders) | 2/943 | 1/929
Chest pain (General disorders) | 21/943 | 15/929
Death (General disorders) | 2/943 | 3/929
Drowning (General disorders) | 2/943 | 1/929
Fatigue (General disorders) | 1/943 | 0/929
General physical health deterioration (General disorders) | 0/943 | 2/929
Hernia (General disorders) | 1/943 | 0/929
Impaired healing (General disorders) | 0/943 | 1/929
Inflammation (General disorders) | 0/943 | 1/929
Malaise (General disorders) | 1/943 | 1/929
Mechanical complication of implant (General disorders) | 0/943 | 1/929
Multi-organ failure (General disorders) | 1/943 | 3/929
Necrosis (General disorders) | 1/943 | 0/929
Non-cardiac chest pain (General disorders) | 5/943 | 3/929
Oedema peripheral (General disorders) | 2/943 | 0/929
Pain (General disorders) | 0/943 | 1/929
Pyrexia (General disorders) | 6/943 | 2/929
Sudden cardiac death (General disorders) | 0/943 | 1/929
Sudden death (General disorders) | 7/943 | 6/929
Ulcer (General disorders) | 1/943 | 0/929
Cholangitis (Hepatobiliary disorders) | 0/943 | 1/929
Cholecystitis (Hepatobiliary disorders) | 2/943 | 3/929
Cholecystitis acute (Hepatobiliary disorders) | 1/943 | 1/929
Cholelithiasis (Hepatobiliary disorders) | 1/943 | 4/929
Gallbladder pain (Hepatobiliary disorders) | 1/943 | 0/929
Hepatic cirrhosis (Hepatobiliary disorders) | 1/943 | 0/929
Hepatic failure (Hepatobiliary disorders) | 0/943 | 1/929
Jaundice (Hepatobiliary disorders) | 0/943 | 1/929
Anaphylactic reaction (Immune system disorders) | 0/943 | 1/929
Corneal graft rejection (Immune system disorders) | 0/943 | 1/929
Secondary immunodeficiency (Immune system disorders) | 1/943 | 0/929
Anal abscess (Infections and infestations) | 0/943 | 1/929
Appendicitis (Infections and infestations) | 1/943 | 1/929
Arthritis bacterial (Infections and infestations) | 1/943 | 1/929
Arthritis infective (Infections and infestations) | 1/943 | 0/929
Bronchitis (Infections and infestations) | 2/943 | 1/929
Bronchopneumonia (Infections and infestations) | 3/943 | 1/929
Cellulitis (Infections and infestations) | 1/943 | 0/929
Chronic sinusitis (Infections and infestations) | 1/943 | 0/929
Chronic tonsillitis (Infections and infestations) | 0/943 | 1/929
Clostridium difficile colitis (Infections and infestations) | 3/943 | 0/929
Cystitis (Infections and infestations) | 1/943 | 1/929
Diverticulitis (Infections and infestations) | 1/943 | 4/929
Endocarditis (Infections and infestations) | 7/943 | 11/929
Endocarditis bacterial (Infections and infestations) | 1/943 | 1/929
Enterococcal sepsis (Infections and infestations) | 0/943 | 1/929
Erysipelas (Infections and infestations) | 2/943 | 6/929
Febrile infection (Infections and infestations) | 1/943 | 0/929
Fungal infection (Infections and infestations) | 0/943 | 1/929
Gangrene (Infections and infestations) | 1/943 | 0/929
Gastroenteritis (Infections and infestations) | 7/943 | 1/929
Groin abscess (Infections and infestations) | 0/943 | 1/929
Haematoma infection (Infections and infestations) | 1/943 | 0/929
Herpes zoster (Infections and infestations) | 1/943 | 0/929
Infection (Infections and infestations) | 2/943 | 3/929
Influenza (Infections and infestations) | 1/943 | 0/929
Intestinal gangrene (Infections and infestations) | 1/943 | 0/929
Klebsiella sepsis (Infections and infestations) | 1/943 | 0/929
Laryngitis (Infections and infestations) | 1/943 | 0/929
Localised infection (Infections and infestations) | 0/943 | 2/929
Lower respiratory tract infection (Infections and infestations) | 2/943 | 3/929
Lung infection (Infections and infestations) | 0/943 | 1/929
Mastoiditis (Infections and infestations) | 1/943 | 0/929
Mediastinitis (Infections and infestations) | 0/943 | 1/929
Meningitis pneumococcal (Infections and infestations) | 0/943 | 1/929
Nasopharyngitis (Infections and infestations) | 0/943 | 1/929
Neuroborreliosis (Infections and infestations) | 0/943 | 1/929
Orchitis (Infections and infestations) | 2/943 | 0/929
Peritonsillitis (Infections and infestations) | 0/943 | 1/929
Pneumonia (Infections and infestations) | 28/943 | 31/929
Pneumonia bacterial (Infections and infestations) | 2/943 | 1/929
Pneumonia streptococcal (Infections and infestations) | 0/943 | 1/929
Post procedural infection (Infections and infestations) | 2/943 | 2/929
Postoperative wound infection (Infections and infestations) | 1/943 | 1/929
Pseudomonas infection (Infections and infestations) | 1/943 | 0/929
Pyelonephritis (Infections and infestations) | 1/943 | 2/929
Pyelonephritis acute (Infections and infestations) | 0/943 | 1/929
Pyothorax (Infections and infestations) | 1/943 | 0/929
Rash pustular (Infections and infestations) | 1/943 | 0/929
Respiratory tract infection (Infections and infestations) | 1/943 | 1/929
Sepsis (Infections and infestations) | 6/943 | 6/929
Sinusitis (Infections and infestations) | 1/943 | 0/929
Skin infection (Infections and infestations) | 0/943 | 1/929
Staphylococcal infection (Infections and infestations) | 0/943 | 1/929
Staphylococcal sepsis (Infections and infestations) | 1/943 | 0/929
Sternitis (Infections and infestations) | 0/943 | 1/929
Streptococcal sepsis (Infections and infestations) | 1/943 | 0/929
Subcutaneous abscess (Infections and infestations) | 1/943 | 0/929
Tooth abscess (Infections and infestations) | 0/943 | 1/929
Tracheobronchitis (Infections and infestations) | 0/943 | 1/929
Upper respiratory tract infection (Infections and infestations) | 0/943 | 2/929
Urinary tract infection (Infections and infestations) | 10/943 | 13/929
Urosepsis (Infections and infestations) | 2/943 | 0/929
Viral infection (Infections and infestations) | 3/943 | 1/929
Wound infection (Infections and infestations) | 1/943 | 1/929
Wound infection staphylococcal (Infections and infestations) | 1/943 | 0/929
Alcohol poisoning (Injury, poisoning and procedural complications) | 1/943 | 0/929
Ankle fracture (Injury, poisoning and procedural complications) | 2/943 | 0/929
Arthropod bite (Injury, poisoning and procedural complications) | 1/943 | 0/929
Asbestosis (Injury, poisoning and procedural complications) | 1/943 | 0/929
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0/943 | 1/929
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0/943 | 1/929
Chest injury (Injury, poisoning and procedural complications) | 1/943 | 0/929
Clavicle fracture (Injury, poisoning and procedural complications) | 0/943 | 1/929
Concussion (Injury, poisoning and procedural complications) | 0/943 | 1/929
Contusion (Injury, poisoning and procedural complications) | 2/943 | 0/929
Device failure (Injury, poisoning and procedural complications) | 1/943 | 0/929
Device occlusion (Injury, poisoning and procedural complications) | 0/943 | 1/929
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1/943 | 2/929
Drug administration error (Injury, poisoning and procedural complications) | 1/943 | 0/929
Drug toxicity (Injury, poisoning and procedural complications) | 1/943 | 0/929
Facial bones fracture (Injury, poisoning and procedural complications) | 1/943 | 0/929
Fall (Injury, poisoning and procedural complications) | 7/943 | 3/929
Femoral neck fracture (Injury, poisoning and procedural complications) | 3/943 | 5/929
Femur fracture (Injury, poisoning and procedural complications) | 2/943 | 6/929
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0/943 | 1/929
Hand fracture (Injury, poisoning and procedural complications) | 1/943 | 1/929
Head injury (Injury, poisoning and procedural complications) | 1/943 | 0/929
Hip fracture (Injury, poisoning and procedural complications) | 4/943 | 4/929
Humerus fracture (Injury, poisoning and procedural complications) | 2/943 | 1/929
Incision site pain (Injury, poisoning and procedural complications) | 0/943 | 1/929
Incisional hernia (Injury, poisoning and procedural complications) | 0/943 | 2/929
Jaw fracture (Injury, poisoning and procedural complications) | 0/943 | 1/929
Joint dislocation (Injury, poisoning and procedural complications) | 1/943 | 1/929
Lower limb fracture (Injury, poisoning and procedural complications) | 1/943 | 0/929
Medical device complication (Injury, poisoning and procedural complications) | 1/943 | 2/929
Meniscus lesion (Injury, poisoning and procedural complications) | 2/943 | 3/929
Multiple fractures (Injury, poisoning and procedural complications) | 1/943 | 0/929
Open wound (Injury, poisoning and procedural complications) | 1/943 | 0/929
Operative haemorrhage (Injury, poisoning and procedural complications) | 0/943 | 1/929
Overdose (Injury, poisoning and procedural complications) | 1/943 | 2/929
Pelvic fracture (Injury, poisoning and procedural complications) | 0/943 | 1/929
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1/943 | 4/929
Postoperative constipation (Injury, poisoning and procedural complications) | 1/943 | 0/929
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1/943 | 0/929
Procedural pain (Injury, poisoning and procedural complications) | 1/943 | 1/929
Procedural site reaction (Injury, poisoning and procedural complications) | 1/943 | 0/929
Pubic rami fracture (Injury, poisoning and procedural complications) | 1/943 | 0/929
Radius fracture (Injury, poisoning and procedural complications) | 2/943 | 1/929
Renal haematoma (Injury, poisoning and procedural complications) | 1/943 | 0/929
Rib fracture (Injury, poisoning and procedural complications) | 2/943 | 3/929
Road traffic accident (Injury, poisoning and procedural complications) | 2/943 | 0/929
Skin laceration (Injury, poisoning and procedural complications) | 1/943 | 1/929
Skull fracture (Injury, poisoning and procedural complications) | 0/943 | 1/929
Snake bite (Injury, poisoning and procedural complications) | 1/943 | 0/929
Spinal fracture (Injury, poisoning and procedural complications) | 1/943 | 1/929
Subdural haematoma (Injury, poisoning and procedural complications) | 1/943 | 0/929
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0/943 | 1/929
Tendon rupture (Injury, poisoning and procedural complications) | 0/943 | 2/929
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0/943 | 1/929
Thermal burn (Injury, poisoning and procedural complications) | 0/943 | 1/929
Tibia fracture (Injury, poisoning and procedural complications) | 1/943 | 0/929
Ulna fracture (Injury, poisoning and procedural complications) | 1/943 | 1/929
Upper limb fracture (Injury, poisoning and procedural complications) | 1/943 | 2/929
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0/943 | 1/929
Wound dehiscence (Injury, poisoning and procedural complications) | 0/943 | 1/929
Wrist fracture (Injury, poisoning and procedural complications) | 1/943 | 0/929
Dehydration (Metabolism and nutrition disorders) | 1/943 | 0/929
Diabetes mellitus (Metabolism and nutrition disorders) | 1/943 | 0/929
Hyperkalaemia (Metabolism and nutrition disorders) | 0/943 | 1/929
Hypokalaemia (Metabolism and nutrition disorders) | 0/943 | 1/929
Hyponatraemia (Metabolism and nutrition disorders) | 1/943 | 1/929
Podagra (Metabolism and nutrition disorders) | 0/943 | 1/929
Arthralgia (Musculoskeletal and connective tissue disorders) | 4/943 | 1/929
Arthritis (Musculoskeletal and connective tissue disorders) | 4/943 | 2/929
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1/943 | 1/929
Arthropathy (Musculoskeletal and connective tissue disorders) | 3/943 | 0/929
Articular calcification (Musculoskeletal and connective tissue disorders) | 0/943 | 1/929
Back pain (Musculoskeletal and connective tissue disorders) | 3/943 | 2/929
Bursitis (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
CREST syndrome (Musculoskeletal and connective tissue disorders) | 0/943 | 2/929
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
Flank pain (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
Foot deformity (Musculoskeletal and connective tissue disorders) | 1/943 | 1/929
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0/943 | 1/929
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4/943 | 0/929
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
Limb deformity (Musculoskeletal and connective tissue disorders) | 0/943 | 1/929
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 0/943 | 1/929
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1/943 | 1/929
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2/943 | 2/929
Myalgia (Musculoskeletal and connective tissue disorders) | 1/943 | 1/929
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0/943 | 1/929
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19/943 | 21/929
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
Osteolysis (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2/943 | 1/929
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/943 | 2/929
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
Periarthritis (Musculoskeletal and connective tissue disorders) | 0/943 | 1/929
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0/943 | 2/929
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1/943 | 1/929
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2/943 | 3/929
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2/943 | 5/929
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/943 | 1/929
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0/943 | 1/929
Synovitis (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1/943 | 0/929
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/943 | 0/929
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 3/929
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9/943 | 4/929
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/943 | 4/929
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 2/929
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8/943 | 2/929
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 1/929
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/943 | 4/929
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 1/929
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 1/929
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 1/929
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 2/929
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 3/929
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/943 | 2/929
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/943 | 2/929
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Metastases to gallbladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/943 | 0/929
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 2/929
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 3/929
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 1/929
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21/943 | 14/929
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 1/929
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 1/929
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/943 | 3/929
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 1/929
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 1/929
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/943 | 1/929
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/943 | 1/929
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 2/929
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/943 | 0/929
Amyotrophic lateral sclerosis (Nervous system disorders) | 0/943 | 1/929
Balance disorder (Nervous system disorders) | 1/943 | 1/929
Carotid artery stenosis (Nervous system disorders) | 0/943 | 1/929
Carotid sinus syndrome (Nervous system disorders) | 1/943 | 0/929
Cerebral infarction (Nervous system disorders) | 2/943 | 1/929
Cerebrovascular accident (Nervous system disorders) | 2/943 | 4/929
Cognitive disorder (Nervous system disorders) | 0/943 | 2/929
Convulsion (Nervous system disorders) | 2/943 | 2/929
Dementia (Nervous system disorders) | 0/943 | 1/929
Dementia Alzheimer's type (Nervous system disorders) | 0/943 | 1/929
Dizziness (Nervous system disorders) | 7/943 | 3/929
Encephalitis (Nervous system disorders) | 1/943 | 0/929
Epilepsy (Nervous system disorders) | 7/943 | 2/929
Facial palsy (Nervous system disorders) | 1/943 | 0/929
Global amnesia (Nervous system disorders) | 1/943 | 0/929
Haemorrhagic stroke (Nervous system disorders) | 1/943 | 0/929
Headache (Nervous system disorders) | 1/943 | 2/929
Hemiparesis (Nervous system disorders) | 1/943 | 0/929
Hypoaesthesia (Nervous system disorders) | 0/943 | 1/929
Intracranial aneurysm (Nervous system disorders) | 0/943 | 1/929
Motor neurone disease (Nervous system disorders) | 1/943 | 0/929
Narcolepsy (Nervous system disorders) | 0/943 | 1/929
Presyncope (Nervous system disorders) | 2/943 | 5/929
Radicular syndrome (Nervous system disorders) | 0/943 | 1/929
Senile dementia (Nervous system disorders) | 0/943 | 1/929
Somnolence (Nervous system disorders) | 1/943 | 0/929
Spinal cord compression (Nervous system disorders) | 0/943 | 1/929
Subarachnoid haemorrhage (Nervous system disorders) | 1/943 | 1/929
Subdural hygroma (Nervous system disorders) | 1/943 | 0/929
Syncope (Nervous system disorders) | 14/943 | 19/929
Syncope vasovagal (Nervous system disorders) | 2/943 | 1/929
Transient ischaemic attack (Nervous system disorders) | 11/943 | 11/929
Anxiety (Psychiatric disorders) | 2/943 | 0/929
Completed suicide (Psychiatric disorders) | 1/943 | 0/929
Confusional state (Psychiatric disorders) | 3/943 | 0/929
Delusional disorder, persecutory type (Psychiatric disorders) | 0/943 | 1/929
Depression (Psychiatric disorders) | 3/943 | 2/929
Major depression (Psychiatric disorders) | 2/943 | 0/929
Mental disorder (Psychiatric disorders) | 0/943 | 1/929
Mental disorder due to a general medical condition (Psychiatric disorders) | 1/943 | 0/929
Panic attack (Psychiatric disorders) | 0/943 | 1/929
Psychosomatic disease (Psychiatric disorders) | 0/943 | 1/929
Anuria (Renal and urinary disorders) | 0/943 | 1/929
Azotaemia (Renal and urinary disorders) | 0/943 | 2/929
Bladder obstruction (Renal and urinary disorders) | 0/943 | 1/929
Calculus bladder (Renal and urinary disorders) | 1/943 | 1/929
Calculus urinary (Renal and urinary disorders) | 2/943 | 2/929
Haematuria (Renal and urinary disorders) | 3/943 | 3/929
Hydronephrosis (Renal and urinary disorders) | 1/943 | 0/929
Nephritis interstitial (Renal and urinary disorders) | 0/943 | 1/929
Nephrolithiasis (Renal and urinary disorders) | 3/943 | 1/929
Renal artery arteriosclerosis (Renal and urinary disorders) | 0/943 | 1/929
Renal failure (Renal and urinary disorders) | 1/943 | 5/929
Renal failure acute (Renal and urinary disorders) | 0/943 | 1/929
Renal impairment (Renal and urinary disorders) | 2/943 | 1/929
Urethral meatus stenosis (Renal and urinary disorders) | 0/943 | 1/929
Urethral stenosis (Renal and urinary disorders) | 0/943 | 1/929
Urinary bladder polyp (Renal and urinary disorders) | 0/943 | 2/929
Urinary incontinence (Renal and urinary disorders) | 1/943 | 0/929
Urinary retention (Renal and urinary disorders) | 3/943 | 4/929
Acquired hydrocele (Reproductive system and breast disorders) | 0/943 | 1/929
Bartholinitis (Reproductive system and breast disorders) | 0/943 | 1/929
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3/943 | 9/929
Cystocele (Reproductive system and breast disorders) | 2/943 | 0/929
Endometrial hyperplasia (Reproductive system and breast disorders) | 0/943 | 1/929
Epididymitis (Reproductive system and breast disorders) | 1/943 | 0/929
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0/943 | 1/929
Ovarian cyst (Reproductive system and breast disorders) | 1/943 | 0/929
Pelvic pain (Reproductive system and breast disorders) | 0/943 | 1/929
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0/943 | 2/929
Prostatism (Reproductive system and breast disorders) | 1/943 | 0/929
Prostatomegaly (Reproductive system and breast disorders) | 1/943 | 0/929
Spermatocele (Reproductive system and breast disorders) | 1/943 | 1/929
Uterine malposition (Reproductive system and breast disorders) | 1/943 | 0/929
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1/943 | 0/929
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 1/943 | 0/929
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3/943 | 5/929
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12/943 | 12/929
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2/943 | 1/929
Eosinophilic pneumonia chronic (Respiratory, thoracic and mediastinal disorders) | 1/943 | 0/929
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9/943 | 1/929
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1/943 | 0/929
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1/943 | 0/929
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0/943 | 1/929
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1/943 | 0/929
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0/943 | 1/929
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9/943 | 7/929
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0/943 | 1/929
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3/943 | 0/929
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 3/943 | 0/929
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2/943 | 4/929
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0/943 | 1/929
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1/943 | 0/929
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3/943 | 4/929
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2/943 | 1/929
Angioedema (Skin and subcutaneous tissue disorders) | 0/943 | 1/929
Dermal cyst (Skin and subcutaneous tissue disorders) | 1/943 | 0/929
Dermatitis (Skin and subcutaneous tissue disorders) | 0/943 | 1/929
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0/943 | 1/929
Eczema (Skin and subcutaneous tissue disorders) | 1/943 | 0/929
Pemphigoid (Skin and subcutaneous tissue disorders) | 1/943 | 0/929
Rash (Skin and subcutaneous tissue disorders) | 1/943 | 1/929
Skin ulcer (Skin and subcutaneous tissue disorders) | 2/943 | 2/929
Urticaria (Skin and subcutaneous tissue disorders) | 0/943 | 1/929
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0/943 | 1/929
Cardiac assistance device user (Social circumstances) | 1/943 | 0/929
Angiodysplasia (Vascular disorders) | 1/943 | 1/929
Aortic aneurysm (Vascular disorders) | 6/943 | 4/929
Aortic dissection (Vascular disorders) | 1/943 | 0/929
Aortic rupture (Vascular disorders) | 0/943 | 1/929
Arteriovenous fistula (Vascular disorders) | 1/943 | 0/929
Bleeding varicose vein (Vascular disorders) | 0/943 | 1/929
Circulatory collapse (Vascular disorders) | 1/943 | 1/929
Deep vein thrombosis (Vascular disorders) | 1/943 | 2/929
Femoral artery aneurysm (Vascular disorders) | 1/943 | 1/929
Haematoma (Vascular disorders) | 3/943 | 3/929
Haemorrhage (Vascular disorders) | 4/943 | 1/929
Hypertension (Vascular disorders) | 0/943 | 3/929
Hypertensive crisis (Vascular disorders) | 2/943 | 2/929
Hypotension (Vascular disorders) | 2/943 | 0/929
Intermittent claudication (Vascular disorders) | 2/943 | 3/929
Orthostatic hypotension (Vascular disorders) | 2/943 | 0/929
Peripheral arterial occlusive disease (Vascular disorders) | 0/943 | 2/929
Phlebitis superficial (Vascular disorders) | 1/943 | 0/929
Raynaud's phenomenon (Vascular disorders) | 0/943 | 1/929
Shock (Vascular disorders) | 1/943 | 0/929
Shock haemorrhagic (Vascular disorders) | 1/943 | 0/929
Thrombophlebitis (Vascular disorders) | 1/943 | 1/929
Varicose vein (Vascular disorders) | 2/943 | 1/929
Vascular occlusion (Vascular disorders) | 0/943 | 1/929
Vascular pseudoaneurysm (Vascular disorders) | 0/943 | 2/929
Venous stasis (Vascular disorders) | 0/943 | 1/929
Venous thrombosis (Vascular disorders) | 2/943 | 1/929
Venous thrombosis limb (Vascular disorders) | 1/943 | 0/929
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | EZ/Simva 10/40 mg | Placebo
Anaemia (Blood and lymphatic system disorders) | 50/943 | 33/929
Angina pectoris (Cardiac disorders) | 36/943 | 44/929
Aortic valve stenosis (Cardiac disorders) | 139/943 | 177/929
Atrial fibrillation (Cardiac disorders) | 88/943 | 113/929
Atrioventricular block first degree (Cardiac disorders) | 23/943 | 11/929
Cardiac failure (Cardiac disorders) | 19/943 | 24/929
Coronary artery disease (Cardiac disorders) | 25/943 | 33/929
Palpitations (Cardiac disorders) | 19/943 | 17/929
Vertigo (Ear and labyrinth disorders) | 27/943 | 28/929
Cataract (Eye disorders) | 22/943 | 33/929
Constipation (Gastrointestinal disorders) | 30/943 | 38/929
Diarrhoea (Gastrointestinal disorders) | 39/943 | 39/929
Dyspepsia (Gastrointestinal disorders) | 23/943 | 16/929
Gastritis (Gastrointestinal disorders) | 22/943 | 19/929
Nausea (Gastrointestinal disorders) | 39/943 | 21/929
Alanine aminotransferase increased (General disorders) | 34/943 | 17/929
Aspartate aminotransferase increased (General disorders) | 38/943 | 15/929
Blood creatine phosphokinase increased (General disorders) | 32/943 | 27/929
Blood glucose increased (General disorders) | 15/943 | 22/929
C-reactive protein increased (General disorders) | 6/943 | 21/929
Gamma-glutamyltransferase increased (General disorders) | 28/943 | 20/929
Haemoglobin decreased (General disorders) | 23/943 | 23/929
Weight decreased (General disorders) | 22/943 | 23/929
Chest pain (General disorders) | 45/943 | 52/929
Fatigue (General disorders) | 43/943 | 41/929
Oedema peripheral (General disorders) | 59/943 | 51/929
Bronchitis (Infections and infestations) | 39/943 | 45/929
Cystitis (Infections and infestations) | 14/943 | 24/929
Influenza (Infections and infestations) | 21/943 | 22/929
Nasopharyngitis (Infections and infestations) | 57/943 | 55/929
Pneumonia (Infections and infestations) | 45/943 | 41/929
Urinary tract infection (Infections and infestations) | 51/943 | 51/929
Diabetes mellitus (Metabolism and nutrition disorders) | 21/943 | 17/929
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0/943 | 19/929
Arthralgia (Musculoskeletal and connective tissue disorders) | 61/943 | 45/929
Back pain (Musculoskeletal and connective tissue disorders) | 56/943 | 48/929
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 19/943 | 39/929
Myalgia (Musculoskeletal and connective tissue disorders) | 41/943 | 51/929
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 29/943 | 39/929
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32/943 | 34/929
Dizziness (Nervous system disorders) | 73/943 | 77/929
Headache (Nervous system disorders) | 26/943 | 32/929
Syncope (Nervous system disorders) | 20/943 | 19/929
Depression (Psychiatric disorders) | 38/943 | 34/929
Insomnia (Psychiatric disorders) | 25/943 | 23/929
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 26/943 | 20/929
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8/943 | 20/929
Cough (Respiratory, thoracic and mediastinal disorders) | 38/943 | 35/929
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 81/943 | 116/929
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 25/943 | 20/929
Eczema (Skin and subcutaneous tissue disorders) | 18/943 | 19/929
Rash (Skin and subcutaneous tissue disorders) | 26/943 | 25/929
Hypertension (Vascular disorders) | 133/943 | 148/929

LIMITATIONS AND CAVEATS:
It is important to note that several of the ischemic outcomes making up the composite ischemic endpoint can occur as a causal consequence of aortic stenosis progression itself, or in association with its standard treatment (aortic valve replacement).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.